CLINICAL TRIAL: NCT06299592
Title: Comparison of Microglial Activation in Severe Asthma and Healthy Controls
Acronym: MAIA-SC
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2023-1626; 1RF1AG082215-01 (NIH); A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison); Protocol Version 7/1/2025 (Other: UW Madison)
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood
  * Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Participants with asthma
  Interventions: Combination Product: PET/MRI using [18F]FEPPA tracer
- Participants without asthma
  Interventions: Combination Product: PET/MRI using [18F]FEPPA tracer

INTERVENTIONS:
Combination Product: PET/MRI using [18F]FEPPA tracer — PET/MRI scans with [18F]FEPPA radiotracer selective for translocator protein (TSPO) binding, which is elevated in activated microglia

SUMMARY:
The goal of this clinical trial is to learn about how asthma influences brain function. The main questions it aims to answer are:

* How airway inflammation in asthma affects the brain; and,
* Whether airway inflammation in asthma is related to symptoms of depression and anxiety

Over the course of 3 visits, participants will:

* Complete questionnaires
* Complete computer tasks
* Undergo allergy skin test and breathing tests
* Give two blood samples
* Give a sputum sample
* Complete brain imaging scans

Researchers will compare results between participants with asthma, and participants who do not have asthma.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Individuals with no health concerns that might affect the outcome of the study
* Age 18-75 years of age
* Ability to tolerate a simulated MRI brain scanning session
* In the opinion of the investigator, capable and willing to grant written informed consent and cooperate with study procedures and requirements
* High-affinity TSPO-binding genotype. Mixed (high/low) binding-affinity genotype may be included at PIs discretion
* For participants with severe asthma:

  * Physician diagnosis of asthma for at least six months prior to screening (can be determined at the discretion of an asthma/allergy physician member of the study team)
  * Severe asthmatics must meet the ATS definition of severe asthma and/or be currently receiving a GINA Step 4 or 5 therapy or daily treatment of 320mcg budesonide. Therapy may include ongoing use of currently approved biologic immunomodulators

Exclusion Criteria:

* Current smoker (defined as more than 0.5 pack per week for the past 6 months and any smoking within two weeks of study procedures) or has a smoking history exceeding 5 pack years within the last 10 years
* Currently receiving allergen immunotherapy unless on stable dose.
* Use of psychotropic medication that might affect function of neurocircuitry implicated in our hypotheses (at the discretion of the PI/Co-I)
* Inability to hold medications detailed in the medication hold schedule
* Needle phobia or claustrophobia
* Major health problems such any of the following in the last 6 months: stroke/TIA, myocardial Infarction, stent placement, or acute coronary syndrome are definitively exclusionary. Decisions regarding other major health problems, such as autoimmune disease, history of carotid stenosis, heart disease, uncontrolled hypertension, lung diseases other than asthma, history of significant arrhythmias, etc. will be based upon the judgement of the PI/Co-I.
* Use of biologic medication that might affect signaling pathways under investigation (at the discretion of the PI/Co-I)
* Pre-existing chronic infectious disease
* Scheduled use of non-selective beta-blockers prior to each study visit.
* Use of an investigational drug within 30 days of entering the study. This criterion will be reviewed on a case by case basis by the PI/Co-I to determine appropriate washout period. Appropriate wash out period may be greater than 30 days depending on the half-life of the investigational drug. Participants may be eligible for study participation after completing the washout period designated by the PI or Co-I (physician only).
* Any MRI incompatibility as determined by most current MRI screening form
* History of a diagnosed bipolar disorder, schizophrenia, or schizoaffective disorder
* History of serious head trauma or seizure disorder (can be included at the discretion of the PI or Co-I)
* Unable, in the judgement of the investigator, to comply with directions and/or tolerate the procedures required for participation in this study
* Pregnant or breast-feeding or has a planned pregnancy during the course of the study
* Any other medical condition or disease that would impact participant safety or data integrity in the opinion of the PI/CO-I

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (age 18-75) with or without severe asthma.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Binding of [18F]-FEPPA | Up to 2 weeks
  A whole-brain voxel-wise t-test will be performed in FMRIB Software Library (FSL) to identify regions where [18F]-FEPPA binding is significantly different between groups.

SECONDARY OUTCOMES:
How activated microglia correspond to immune biomarkers in lung and blood | Up to 2 weeks
  Whole-brain voxel-wise regressions in FSL will test the relationship between [18F]-FEPPA binding and cytokine levels
Relationship between activated microglia and cognitive function | Up to 2 weeks
  whole-brain voxel-wise regressions in FSL will test the relationship between [18F]-FEPPA binding and cognitive function
Relationship between activated microglia and psychological symptoms | Up to 2 weeks
  whole-brain voxel-wise regressions in FSL will test the relationship between [18F]-FEPPA binding and psychological symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Rosenkranz, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Center for Healthy Minds, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No